CLINICAL TRIAL: NCT05597475
Title: Visualizing Beta Cells in Patients With Hyperinsulinemic Hypoglycemia After Bariatric Surgery
Brief Title: GLP1R-imaging in Post-RYGB Hypoglycemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Principal Investigator, Laura Deden, Principal Investigator, Rijnstate Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NL51854.091.15
Record Dates: First submitted 2020-10-05; First posted 2022-10-28 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Obesity; Hypoglycemia Post Gastric Bypass Surgery; Hyperinsulinemic Hypoglycemia
MeSH Terms: conditions — Obesity; Congenital Hyperinsulinism

ARMS (2):
- Patients (Other): Patients with hypoglycemia
  Interventions: Diagnostic Test: GLP-1R PET
- Controls (Other): Patients without post-bariatric hypoglycemia
  Interventions: Diagnostic Test: GLP-1R PET

INTERVENTIONS:
Diagnostic Test: GLP-1R PET — Beta cell function (tests) and measure for beta cell mass (PET)
  Other Names: Meal tolerance test; Arginine stimulation test

SUMMARY:
In order to evaluate the difference in beta cell mass in patients with and without hyperinsulinemic hypoglycemia after Roux en Y gastric bypass (RYGB) investigators aim to compare quantitative PET imaging of the pancreas between these patient groups.

These highly relevant data will provide investigators with more information on the possible role of beta cell mass in the mechanisms of hyperinsulinemic hypoglycemia bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent

Patients:

- Persisting hyperinsulinemic hypoglycemia after a low-carbohydrate diet and/or insulin suppressive medication for one year.

Controls:

* RYGB at least 2 years ago
* Normal glucose levels before and after RYGB (fasting glucose between 4 and 6 mmol/l or HbA1c between 20 and 42 mmol/mol)
* Score ≤ 7 on Sigstad's scoring system (Table 1)
* Hypoglycemia excluded by 14-day continuous glucose monitoring
* Individual matched to HH group on age (± 5 years), sex and BMI at time of inclusion (± 2 kg/m2)

Exclusion Criteria:

* Anti-diabetic medication in the past 6 months
* Treatment with synthetic Exendin (Exenatide, Byetta®) or Dipeptidyl-Peptidase IV inhibitors in the past six months.
* Known liver failure or serum liver values over 2 times normal value at the time of standard laboratory assessment. Normal values of total bilirubin, γ-GT, ASAT and albumin are <21 μmol, <40 U/l, <30 U/l and 35-50 g/l respectively
* Pregnancy or the wish to become pregnant within 6 months
* Breast feeding
* Kidney failure, i.e. calculated creatinine clearance below 40 ml/min
* Age < 18 years
* No signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Pancreatic uptake of 68Ga-NODAGA-exendin-4 | baseline

SECONDARY OUTCOMES:
Beta cell function | baseline
  Measured as total insulin during MTT and insulin peak during arginine test

CONTACTS AND LOCATIONS:
Locations (1):
- Rijnstate hospital, Arnhem, Netherlands